CLINICAL TRIAL: NCT01778153
Title: Effectiveness of Equinox Fitness Club's Personal Coaching Method Versus Self-Directed Exercise Training on Increasing Lean Body Mass in Men Aged 30-44 Years of Age
Brief Title: Equinox Personal Coaching Versus Self-Directed Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Equinox Fitness Centers (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Equinox Study
Record Dates: First submitted 2011-12-16; First posted 2013-01-29 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Physical Fitness
Keywords: Fitness training; Personal training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Equinox Personal Coaching (Experimental): Participants assigned the Coached group will receive up to 36 sessions about three times a week, consisting of both strength and aerobic exercises, through a program designed by Equinox Fitness Centers.
  Interventions: Behavioral: Equinox Personal Coaching
- Self-directed exercise training (No Intervention): Participants in the Self-directed group will receive general exercise training advice as any member of the fitness club would, and will record the details of their exercise in log sheets. They will be asked to continue their usual exercise routine.

INTERVENTIONS:
Behavioral: Equinox Personal Coaching — Specially designed strength and aerobic exercise training program that consists of 36 sessions over 12 weeks.
  Arms: Equinox Personal Coaching

SUMMARY:
The purpose of this study is to compare the Equinox Personal Coaching exercise training method to self-directed exercise training in helping subjects become more fit. Men between 30 and 44 years of age who exercise on a regular basis and are interested in receiving Equinox personal training will be invited to participate. The investigators will enroll 36 subjects at University of California, Los Angeles (UCLA), the only site. The hypothesis of this study is that subjects randomized to the Personal Coaching Method will result in significantly greater lean mass accrual than those randomized to self-directed training over the 12 weeks of the study.

Subjects will have 2 Baseline visits over 1 week, then be randomized to receive either Coached training or self-training, which they will do for 12 weeks, then complete two End of Study visits over the final week. Visits 1 and 3 include questionnaires, skinfold fat/lean body mass measurements, and strength and aerobic performance tests, and will take place at Equinox. Visits 2 and 4 include a DEXA scan and ECG, which will take place at UCLA.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 30-44 years
* Body mass index less than 30 kg/m2.
* Currently exercising with or without coaching more than 4 days but less than 8 days per month for the past three months (Equinox Motivated or Super Motivated categories);
* Willing to commit to 12 weeks of thrice weekly training at the Century City Equinox club with or without an Equinox coach.

Exclusion Criteria:

* Over age 44
* Musculoskeletal conditions limiting participation
* Unstable cardiovascular, pulmonary, metabolic, or other disorders that would preclude high intensity exercise training.
* Abnormal ECG at Screening that indicates the subject is not healthy enough for maximal exercise in the opinion of the principal investigator
* Family history of sudden death associated with exercise, based on self-report

Ages: 30 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in lean body mass | Baseline and 4 months
  Change in lean body mass (LBM) as measured by dual-energy x-ray absorptiometry (DEXA)

SECONDARY OUTCOMES:
Change in muscle strength | Baseline and 4 months
  Changes in muscle strength in the upper and lower extremities as assessed with standard one-repetition maximum tests for the chest press and leg press exercises, respectively
Change in aerobic performance | Baseline and 4 months
  Aerobic performance as assessed using a symptom-limited, treadmill ramp protocol.
Changes in ventilation and respiratory gas exchange | Baseline and 4 months
  Measures of ventilation and respiratory gas exchange including changes in maximum oxygen uptake, the metabolic (lactate) threshold, and other parameters of aerobic, cardiovascular, and ventilatory fitness.
Change in quality of life | Baseline and 4 months
  A quality of life scale will also used to determine participant's satisfaction with their training and its result.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher B Cooper, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA David Geffen School of Medicine, Los Angeles, California, United States

REFERENCES:
- [Result] Storer TW, Dolezal BA, Berenc MN, Timmins JE, Cooper CB. Effect of supervised, periodized exercise training vs. self-directed training on lean body mass and other fitness variables in health club members. J Strength Cond Res. 2014 Jul;28(7):1995-2006. doi: 10.1519/JSC.0000000000000331. PMID 24276303